CLINICAL TRIAL: NCT01626820
Title: Immunogenicity and Safety Study of GSK Biologicals' Trivalent Split Virion Influenza Vaccine (GSK1536489A) Fluviral® (2012/2013 Season) in Adults Aged 18 Years and Older
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Fluviral® (2012/2013 Season) in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 116664
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2016-08

CONDITIONS: Influenza
Keywords: Immunogenicity; Influenza; Safety; Adults; Fluviral
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (2):
- Fluviral Adults Group (Experimental): Subjects 18-60 years of age received 1 dose of Fluviral® vaccine, administered intramuscularly in the deltoid of the non-dominant arm, at Day 0.
  Interventions: Biological: Fluviral®
- Fluviral Elderly Group (Experimental): Subjects above 60 years of age received 1 dose of Fluviral® vaccine, administered intramuscularly in the deltoid of the non-dominant arm, at Day 0.
  Interventions: Biological: Fluviral®

INTERVENTIONS:
Biological: Fluviral® — 1 dose administered intramuscularly in deltoid region of non-dominant arm at Day 0

SUMMARY:
This study is designed to test the immunogenicity in terms of Hemagglutination Inhibition (HI) antibodies against each of the three vaccine influenza strains and reactogenicity and safety of Fluviral® containing the influenza strains recommended for the 2012-2013 season.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female 18 years of age and older at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Administration of any influenza vaccine within 6 months preceding the study start or planned use of such vaccines during the study period.
* Administration of any other vaccine(s) within 30 days prior to study enrolment or during the study period.
* Clinically or virologically confirmed influenza infection within the six months preceding the study vaccination.
* Acute disease and/or fever at the time of enrolment.
* Significant acute or chronic, uncontrolled medical or psychiatric or neurological illness.
* Any confirmed or suspected immunosuppressive or immunodeficient condition.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Insulin-dependent diabetes mellitus.
* Presence of blood dyscrasias, including hemoglobinopathies and myelo- or lymphoproliferative disorder.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* A history of any demyelinating disease including Multiple Sclerosis and Guillain-Barré syndrome.
* History of chronic alcohol abuse and/or drug abuse as deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Any significant disorder of coagulation that increases the risk of intramuscular injections or treatment with coumadin derivatives or heparin. Persons receiving prophylactic antiplatelet medications, e.g. low-dose aspirin, and without a clinically-apparent bleeding tendency are eligible.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Any known or suspected allergy to any constituent of Fluviral® and/or a history of anaphylactic type reaction to consumption of eggs, and/or reactions to products containing mercury.
* A history of severe adverse reaction to a previous influenza vaccination.
* Pregnant and/or lactating/nursing female.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-07-19; Primary Completion 2012-08-10 (Actual); Study Completion 2012-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 116664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116664 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At least 50% of the subjects in Fluviral Adults and Fluviral Elderly Groups had not been previously immunized with influenza vaccine in the 2011/2012 season.
Groups:
- Fluviral Elderly Group: Subjects above 60 years of age received 1 dose of Fluviral® vaccine, administered intramuscularly in the deltoid of the non-dominant arm at Day 0
Period: Overall Study
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Started | 56 | 57
Completed | 56 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.80 (12.32) | 68.30 (5.28) | 54.18 (17.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers, Against Each of the Vaccine Influenza Virus Strains.
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine influenza strains included Flu A/CAL/7/09 (H1N1), Flu A/Victoria/361/11 (H3N2) and Flu B/Hubei-Wujiagang/158/09 (Yamagata) antigens.
Time Frame: At Day 0 and Day 21
Population: Analysis was performed on According To Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Number analyzed (Participants) | 56 | 56
Titer
  [H1N1 strain, Day 0] | 84.03 [56.69 to 124.57] | 40.48 [27.97 to 58.58]
  [H1N1 strain, Day 21] | 306.51 [237.33 to 395.86] | 159.02 [116.82 to 216.46]
  [H3N2 strain, Day 0] | 24.82 [17.10 to 36.04] | 37.33 [25.78 to 54.06]
  [H3N2 strain, Day 21] | 151.32 [109.35 to 209.39] | 167.04 [117.38 to 237.71]
  [Yamagata strain, Day 0] | 82.50 [60.43 to 112.63] | 65.58 [52.23 to 82.35]
  [Yamagata strain, Day 21] | 328.03 [253.70 to 424.14] | 234.79 [187.46 to 294.06]

2. Primary Outcome: Number of Subjects Seroprotected for HI Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a subject with serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The influenza vaccine strains included Flu A/CAL/7/09 (H1N1), Flu A/Victoria/361/11 (H3N2) and Flu B/Hubei-Wujiagang/158/09 (Yamagata) antigens.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Number analyzed (Participants) | 56 | 56
Subjects
  [H1N1 strain, Day 0] | 43 | 31
  [H1N1 strain, Day 21] | 56 | 53
  [H3N2 strain, Day 0] | 25 | 32
  [H3N2 strain, Day 21] | 51 | 51
  [Yamagata strain, Day 0] | 47 | 46
  [Yamagata strain, Day 21] | 56 | 56

3. Primary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine influenza strains included Flu A/CAL/7/09 (H1N1), Flu A/Victoria/361/11 (H3N2) and Flu B/Hubei-Wujiagang/158/09 (Yamagata) antigens.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Number analyzed (Participants) | 56 | 56
Subjects
  [H1N1 strain] | 22 | 22
  [H3N2 strain] | 27 | 23
  [Yamagata strain] | 26 | 27

4. Primary Outcome: Mean Geometric Increase (MGI) for HI Antibody Titer Against Each of the Three Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination (Day 21) compared to pre-vaccination (Day 0).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Number analyzed (Participants) | 56 | 56
Fold increase
  [H1N1 strain] | 3.6 [2.5 to 5.4] | 3.9 [2.7 to 5.7]
  [H3N2 strain] | 6.1 [4.0 to 9.4] | 4.5 [3.0 to 6.8]
  [Yamagata strain] | 4.0 [2.9 to 5.5] | 3.6 [2.7 to 4.7]

5. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were ecchymosis, induration, pain, redness and swelling. Any was defined as occurrence of any specified solicited local symptoms reported irrespective of intensity grade. Grade 3 pain was defined as considerable pain that prevented normal everyday activities. Grade 3 ecchymosis, induration, redness and swelling were defined as ecchymosis, induration, redness and swelling above 100 millimeters (mm).
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort which included all subjects with a documented vaccine administration and symptom sheet completed.
Measure: Number; unit: Subjects
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Number analyzed (Participants) | 56 | 57
Subjects
  Any Ecchymosis | 0 | 0
  Grade 3 Ecchymosis | 0 | 0
  Any Induration | 0 | 0
  Grade 3 Induration | 0 | 0
  Any Pain | 41 | 12
  Grade 3 Pain | 0 | 0
  Any Redness | 0 | 1
  Grade 3 Redness | 0 | 0
  Any Swelling | 0 | 0
  Grade 3 Swelling | 0 | 0

6. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, sweating and fever [oral temperature ≥38.0 degrees Celsius (°C)]. Gastrointestinal symptoms included nausea, vomiting, diarrhea and/or abdominal pain. Any =occurrence of any specified solicited general symptoms reported irrespective of intensity grade or relationship to vaccination, Any fever = oral temperature ≥38.0 degrees Celsius (°C). Grade 3 symptoms = symptoms that prevented normal activities. Grade 3 fever = oral temperature ≥39.0°C. Related = symptoms considered by the investigator to have a causal relationship to vaccination
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Analysis was performed on theTotal Vaccinated cohort which included all subjects with a documented vaccine administration and symptom sheet completed
Measure: Number; unit: Subjects
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Number analyzed (Participants) | 56 | 57
Subjects
  Any Arthralgia | 2 | 2
  Grade 3 Arthralgia | 0 | 0
  Related Arthralgia | 2 | 2
  Any Fatigue | 8 | 7
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 8 | 7
  Any Gastrointestinal symptoms | 3 | 0
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 3 | 0
  Any Headache | 10 | 2
  Grade 3 Headache | 0 | 0
  Related Headache | 10 | 2
  Any Myalgia | 8 | 4
  Grade 3 Myalgia | 0 | 0
  Related Myalgia | 8 | 4
  Any Shivering | 1 | 0
  Grade 3 Shivering | 0 | 0
  Related Shivering | 1 | 0
  Any Sweating | 1 | 0
  Grade 3 Sweating | 0 | 0
  Related Sweating | 1 | 0
  Any Fever | 0 | 0
  Grade 3 Fever | 0 | 0
  Related Fever | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 21-day (Days 0-20) post-vaccination period.
Population: Analysis was performed on the Total Vaccinated cohort which included all subjects with a documented vaccine administration.
Measure: Number; unit: Subjects
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Number analyzed (Participants) | 56 | 57
Subjects | 11 | 5

8. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 - Day 20 after vaccination).
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Number analyzed (Participants) | 56 | 57
Subjects
  Any SAE(s) | 0 | 0
  Related SAE(s) | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events:During the entire study period i.e. Days 0-20 after vaccination; Solicited local and general symptoms: During the 4-day (Days 0-3) post-vaccination period; Unsolicited symptoms: During the 21-day (Days 0-20) post-vaccination period.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | Fluviral Adults Group | Fluviral Elderly Group
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/57
Other Adverse Events (participants affected / at risk) | 43/56 | 18/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluviral Adults Group (N=56) | Fluviral Elderly Group (N=57)
Fatigue (General disorders) | 8 | 7
Gastointestinal symptoms (General disorders) | 3 | 0
Headache (General disorders) | 10 | 2
Myalgia (General disorders) | 8 | 4
Pain (General disorders) | 41 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.